CLINICAL TRIAL: NCT00097669
Title: VITATOPS - A Study of VITAmins TO Prevent Stroke
Brief Title: VITATOPS: A Study of VITAmins TO Prevent Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VITATOPS (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other); National Heart Foundation, Australia (Other); Medical Health Research Infrastructure Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ec550
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2014-01

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: VITATOPS; stroke; prevention; multivitamins; homocysteine
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active VITATOPS Tablet (folic acid 2mg, B6 25mg , B12 500ug) (Active Comparator): Active Treatment Arm: VITATOPS study tablet (folate 2 mg, B6 25 mg, B12 500 ug). Taken daily for the duration of the study.
  Interventions: Drug: Active VITATOPS Tablet (folic acid 2mg, B6 25mg , B12 500ug) or placebo
- Placebo Tablet (Placebo Comparator): Placebo Treatment Arm: The placebo tablet will have the same appearance, taste and texture as the vitamin preparation and contains excipients, coating and coating aids.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Active VITATOPS Tablet (folic acid 2mg, B6 25mg , B12 500ug) or placebo — multivitamin
  Other Names: VITATOPS study tablet
  Arms: Active VITATOPS Tablet (folic acid 2mg, B6 25mg , B12 500ug)
Other: Placebo
  Arms: Placebo Tablet

SUMMARY:
The VITATOPS study is a multi-center, randomized, double blind, placebo-controlled secondary stroke prevention trial to determine whether the addition of vitamin supplements (B12 500 ug, B6 25 mg, Folate 2 mg) to best medical/surgical management (including modification of risk factors) will reduce the combined incidence of recurrent vascular events (stroke, myocardial infarction) and vascular death in patients with recent stroke or transient ischemic attack (TIA). All patients presenting to one of the participating neurologists or general physicians within seven months of stroke (ischemic or hemorrhagic) or TIA (eye or brain) are eligible for this trial. Eligible patients will be randomized in a double-blind fashion to receive multi-vitamins or placebo, 1 tablet daily. The primary outcome event is the composite event "stroke, myocardial infarction, or death from any vascular cause", whichever occurs first. Our target is to recruit a total of 8,000 patients over the next two years with a median follow-up of 2.5 years. Recruitment to the trial began in November 1998 and is planned to continue until December 2005. We aim to complete final follow-up by the end of 2006. However, the Steering Committee will be flexible in dictating the need for ongoing recruitment and continuing follow-up, depending on the overall rate of the primary outcome event in the entire cohort at each interim analysis.

DETAILED DESCRIPTION:
Background: Epidemiological studies suggest that raised plasma concentrations of total homocysteine (tHcy) may be a common, causal and treatable risk factor for atherothromboembolic ischemic stroke, dementia and depression. Although tHcy can be lowered effectively with small doses of folic acid, vitamin B12 and vitamin B6, it is not known whether lowering tHcy, by means of multivitamin therapy, can prevent stroke and other major atherothromboembolic vascular events, dementia and depression.

Purpose: To determine whether vitamin supplements (folic acid 2 mg, B6 25 mg, B12 500 ug) reduce the risk of stroke, other serious vascular events, dementia and depression in patients with recent stroke or transient ischemic attacks of the brain or eye (TIA).

Methods: An international, multi-center, randomized, double-blind, placebo-controlled clinical trial.

Subjects: Patients with stroke or TIA in the previous 7 months.

Primary outcome measure: Non-fatal stroke, non-fatal myocardial infarction, or death due to vascular causes.

Secondary outcome measures: TIA, Revascularisation procedures, Dementia, Depression.

Sample size calculation: To reliably identify a 15% reduction in relative risk of the primary outcome event from 8% to 6.8% per year with an alpha of 0.05 and power of 80%, 8,000 patients need to be randomized and followed-up for an average of two years.

Current progress: As of November, 2004, more than 4,400 patients have been randomized in 73 centers in 19 countries in five continents: Australia, Austria, Belgium, Brazil, Hong Kong, Italy, Malaysia, Moldova, Netherlands, New Zealand, Pakistan, Philippines, Portugal, Republic of Georgia, Serbia & Monte Negro, Singapore, Sri Lanka, United Kingdom, and United States.

VITATOPS aims to recruit and follow up 8,000 patients between 2000 and 2006, and provide a reliable estimate of the safety and effectiveness of dietary supplementation with folic acid, vitamin B12, and vitamin B6 in reducing recurrent serious vascular events, dementia and depression among a wide range of patients with stroke and TIA.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within seven months of stroke (ischemic or hemorrhagic) or TIA
* Agree to take study medication
* Be geographically accessible for follow-up
* Provide written informed consent

Exclusion Criteria:

* Taking folic acid or B6 on medical advice
* Use of vitamin supplements containing folate, B6 or B12 (unless patient agrees to take study medication instead of the vitamin supplements which they usually take)
* Taking Methotrexate for any reason
* Pregnancy or women of child-bearing potential who are at risk of pregnancy
* Limited life expectancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8164 (Actual)
Dates: Start 1998-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Hankey, MBBS/MD, Principal Investigator — Royal Perth Hospital / University of Western Australia; Ross Baker, MBBS/BMedSc, Study Director — Royal Perth Hospital; John Eikelboom, MBBS/FRACP, Study Director — Royal Perth Hospital; Konrad Jamrozik, MBBS, Study Director — The University of Queensland; Frank van Bockxmeer, BSc/PhD, Study Director — Royal Perth Hospital; Siobhan Hickling, BSc/MPH, Study Director — The University of Western Australia; Anna Gelavis, BPharm, Study Director — Royal Perth Hospital
Locations (111):
- United States (4):
  - JFK Hospital / Seton Hall University, New York, New York
  - Abington Memorial Hospital, Abington, Pennsylvania
  - South Carolina VA Hospital, Columbia, South Carolina
  - University of South Carolina, Columbia, South Carolina
- Australia (16):
  - Central Coast Neuroscience Research, Gosford
  - Bankstown Hospital, New South Wales
  - John Hunter Hospital, New South Wales
  - Liverpool Hospital, New South Wales
  - Royal Perth Hospital, Perth
  - Greenslopes Hospital, Queensland
  - Nambour Hospital, Queensland
  - Flinders & Griffiths, South Australia
  - Royal Hobart Hospital, Tasmania
  - Alfred Hospital, Victoria
  - Beleura & Frankston Hospital, Victoria
  - Box Hill Hospital, Victoria
  - National Stroke Research Institute - Austin Health, Victoria
  - Fremantle Hospital, Western Australia
  - Joondalup Hospital, Western Australia
  - Sir Charles Gairdner Hospital, Western Australia
- Karl-Franzens University Graz, Graz, Austria
- Algemeen Ziekenhuis Sint-Jan Autonome Verzorgingsinstelling, Bruges, Belgium
- Universidade Federal Fluminense & Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil
- Sarajishvili Institute of Neurology and Neurosurgery, Tbilisi, Georgia
- Hong Kong (2):
  - Queen Mary Hospital, Pokfulam
  - Prince of Wales Hospital, Shatin
- India (23):
  - Rajah Muthaiah Medical College, Annāmalainagar
  - St John's Medical College Hospital, Bangalore
  - SP Medical College, Bikaner
  - Baby Memorial Hospital, Calicut
  - KS Hospital, Chennai
  - Care Hopstial, Hyderabad
  - Mahaveer Hospital & Research Centre, Hyderabad
  - Mediciti Hospital, Hyderabad
  - MGM Medical College & MY Hospital, Indore
  - Monilek Hospital, Jaipur
  - Amrita Institute of Medical Science, Kochi
  - Centauri, The Albert Road Clinic, Kolkata
  - CSMMU, Lucknow
  - Christian Medical College & Hospital, Ludhiana
  - G.B. Pant Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Sadhbavana Medical & Heart Institute, Patiaala
  - Railway Hospital, Perambūr
  - Poona Hospital, Pune
  - Ruby Hall Clinic, Pune
  - Neurocenter, Trichy
  - Care Hospital, Visakhapatnam
  - Mahatma Gandhi Institute, Wardha
- Italy (7):
  - Spedali Civili Di Brescia, Brescia
  - Ospedale di Circolo de Busto Arsizio, Busto Arsizio
  - Ospedale di Macerata, Macerata
  - IRCCS Fondazione Istituto Neurologico C Mondino, Pavia
  - Perugia Stroke Service & Citta Della Peive, Perugia
  - University of Perugia, Perugia
  - Ospedale R Guzzardi, Vittoria
- Malaysia (2):
  - Hospital Universiti Sains Malaysia, Kelantan
  - University of Malaya Medical Centre, Kuala Lumpur
- City Emergency Hospital, Chishinau, Moldova
- Netherlands (3):
  - Slotervaartziekenhuis, Amsterdam
  - Oosterscheldeziekenhuis, Goes
  - University Medical Center Utrecht, Utrecht
- New Zealand (5):
  - Auckland Hospital, Auckland
  - Hawkes Bay Hospital, Hastings
  - Palmerston North Hospital, Palmerston North
  - North Shore Hospital, Takapuna
  - Wellington Hospital, Wellington South
- Pakistan (5):
  - KRL University, Islamabad
  - Pakistan Institute of Medical Sciences, Islamabad
  - DUHS - Civil Hospital, Karachi
  - DUHS - Jinnah Hospital, Karachi
  - POF Hospital Wah Cantt., Wah Cantt
- Philippines (8):
  - Cagayan de Oro Medical Center, Cebu City
  - Cebu Doctor's Hospital, Cebu City
  - Cebu Velez General Hospital/ Visayas Comm. Medical Center, Cebu City
  - Chong Hua Hospital, Cebu City
  - Vicente Sotto Memorial Hospital, Cebu City
  - Cagayan Valley Medical Center, East Santiago City
  - Jose R Reyes Memorial Medical Centre, Manila
  - University Santo Tomas Hospital, Manila
- Portugal (4):
  - Hospital Visconde de Salreu, Estarreja
  - Hospital de Santa Maria, Lisbon
  - Hospital Distrital de Oliverira de Azemeis, Oliveira de Azeméis
  - Hospital Geral de Santo Antonio, Porto
- University of Novi Sad - Neurology & Neurosurgery, Novisad, Serbia
- Singapore General Hospital, Singapore, Singapore
- Sri Lanka (2):
  - National Hospital of Sri Lanka, Colombo
  - University of Kelaniya, Ragama
- United Kingdom (23):
  - University Hospital of North Staffordshire, Stoke-on-Trent, Shaffordshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Redbridge Health Care, Barking
  - Barnsley District Hospital, Barnsley
  - The Royal Victoria Hospital, Belfast
  - Bronglais General Hospital, Ceredigion
  - Western General Hospital, Edinburgh, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - Western Infirmary, Glasgow
  - St Luke's Hospital, Huddersfield
  - William Harvey Hospital, Kent
  - University Hospital Aintree, Liverpool
  - Altnagelvin Hospital, Londonderry
  - Luton and Dunstable Hospital, Luton
  - Royal Victoria Infirmary, Newcastle, Newcastle
  - North Tyneside District General Hospital, North Shields
  - Nottingham City Hospital, Nottingham
  - St Mary's Paddington Hospital, Paddington
  - Rotherham General Hospital, Rotherham
  - Stirling Royal Infirmary, Stirling
  - Stepping Hill Hospital, Stockport
  - Musgrove Park Hosptial, Taunton
  - Torbay Hospital, Torquay

REFERENCES:
- [Derived] Gommans J, Yi Q, Eikelboom JW, Hankey GJ, Chen C, Rodgers H; VITATOPS trial study group. The effect of homocysteine-lowering with B-vitamins on osteoporotic fractures in patients with cerebrovascular disease: substudy of VITATOPS, a randomised placebo-controlled trial. BMC Geriatr. 2013 Sep 3;13:88. doi: 10.1186/1471-2318-13-88. PMID 24004645
- [Derived] Hankey GJ, Ford AH, Yi Q, Eikelboom JW, Lees KR, Chen C, Xavier D, Navarro JC, Ranawaka UK, Uddin W, Ricci S, Gommans J, Schmidt R, Almeida OP, van Bockxmeer FM; VITATOPS Trial Study Group. Effect of B vitamins and lowering homocysteine on cognitive impairment in patients with previous stroke or transient ischemic attack: a prespecified secondary analysis of a randomized, placebo-controlled trial and meta-analysis. Stroke. 2013 Aug;44(8):2232-9. doi: 10.1161/STROKEAHA.113.001886. Epub 2013 Jun 13. PMID 23765945
- [Derived] Cavalieri M, Schmidt R, Chen C, Mok V, de Freitas GR, Song S, Yi Q, Ropele S, Grazer A, Homayoon N, Enzinger C, Loh K, Wong KS, Wong A, Xiong Y, Chang HM, Wong MC, Fazekas F, Eikelboom JW, Hankey GJ; VITATOPS Trial Study Group. B vitamins and magnetic resonance imaging-detected ischemic brain lesions in patients with recent transient ischemic attack or stroke: the VITAmins TO Prevent Stroke (VITATOPS) MRI-substudy. Stroke. 2012 Dec;43(12):3266-70. doi: 10.1161/STROKEAHA.112.665703. Epub 2012 Oct 23. PMID 23093615
- [Derived] Hankey GJ, Eikelboom JW, Yi Q, Lees KR, Chen C, Xavier D, Navarro JC, Ranawaka UK, Uddin W, Ricci S, Gommans J, Schmidt R; VITATOPS trial study group. Antiplatelet therapy and the effects of B vitamins in patients with previous stroke or transient ischaemic attack: a post-hoc subanalysis of VITATOPS, a randomised, placebo-controlled trial. Lancet Neurol. 2012 Jun;11(6):512-20. doi: 10.1016/S1474-4422(12)70091-1. Epub 2012 May 2. PMID 22554931
- [Derived] Hankey GJ, Eikelboom JW, Yi Q, Lees KR, Chen C, Xavier D, Navarro JC, Ranawaka UK, Uddin W, Ricci S, Gommans J, Schmidt R; VITAmins TO Prevent Stroke (VITATOPS) Trial Study Group. Treatment with B vitamins and incidence of cancer in patients with previous stroke or transient ischemic attack: results of a randomized placebo-controlled trial. Stroke. 2012 Jun;43(6):1572-7. doi: 10.1161/STROKEAHA.111.641613. Epub 2012 Apr 3. PMID 22474057
- [Derived] Almeida OP, Marsh K, Alfonso H, Flicker L, Davis TM, Hankey GJ. B-vitamins reduce the long-term risk of depression after stroke: The VITATOPS-DEP trial. Ann Neurol. 2010 Oct;68(4):503-10. doi: 10.1002/ana.22189. PMID 20976769
- [Derived] VITATOPS Trial Study Group. B vitamins in patients with recent transient ischaemic attack or stroke in the VITAmins TO Prevent Stroke (VITATOPS) trial: a randomised, double-blind, parallel, placebo-controlled trial. Lancet Neurol. 2010 Sep;9(9):855-65. doi: 10.1016/S1474-4422(10)70187-3. Epub 2010 Aug 3. PMID 20688574
- [Derived] VITATOPS Trial Study Group; Hankey GJ, Algra A, Chen C, Wong MC, Cheung R, Wong L, Divjak I, Ferro J, de Freitas G, Gommans J, Groppa S, Hill M, Spence D, Lees K, Lisheng L, Navarro J, Ranawaka U, Ricci S, Schmidt R, Slivka A, Tan K, Tsiskaridze A, Uddin W, Vanhooren G, Xavier D, Armitage J, Hobbs M, Le M, Sudlow C, Wheatley K, Yi Q, Bulder M, Eikelboom JW, Hankey GJ, Ho WK, Jamrozik K, Klijn K, Koedam E, Langton P, Nijboer E, Tuch P, Pizzi J, Tang M, Antenucci M, Chew Y, Chinnery D, Cockayne C, Loh K, McMullin L, Smith F, Schmidt R, Chen C, Wong MC, de Freitas G, Hankey GJ, Loh K, Song S. VITATOPS, the VITAmins TO prevent stroke trial: rationale and design of a randomised trial of B-vitamin therapy in patients with recent transient ischaemic attack or stroke (NCT00097669) (ISRCTN74743444). Int J Stroke. 2007 May;2(2):144-50. doi: 10.1111/j.1747-4949.2007.00111.x. PMID 18705976
- See also: National Heart Foundation — http://www.heartfoundation.com.au/
- See also: Stroke Society of Australasia Inc. — http://www.strokesociety.com.au/

RESULTS

PARTICIPANT FLOW:
Groups:
- Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug): Active Treatment Arm: VITATOPS study tablet (folate 2 mg, B6 25 mg, B12 500 ug). Taken daily for the duration of the study.
  Active VITATOPS Tablet (folic acid 2mg, B6 25mg , B12 500ug): multivitamin
Period: Overall Study
Arm/Group | Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug) | Placebo Tablet
Started | 4089 | 4075
Completed | 4089 | 4075
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug) | Placebo Tablet | Total
Number analyzed (Participants) | 4089 | 4075 | 8164
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (12.6) | 62.6 (12.4) | 62.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1475 | 1471 | 2946
  Male | 2614 | 2604 | 5218
Functional severity of qualifying stroke [Number; unit: participants] — Oxford Handicap Score (<3 = functionally independent; 3-5= functional dependent on help)
  participants
    Independent (Oxford handicap score 0-3) | 3035 | 3024 | 6059
    Dependent (Oxford handicap score 3,4 or 5) | 951 | 943 | 1894
past history of stroke, prior to qualifying stroke or transient ischemic attack (TIA) [Number; unit: participants] — This measure refers to the number of randomised patients who had a history of a previous stroke, prior to the stroke or transient ischemic attack (TIA) that qualified them for entry into the trial.
  participants | 624 | 658 | 1282
laboratory results for fasting homocysteine [Mean (Standard Deviation); unit: micromoles per liter] — Fasting blood homocysteine concentrations were measured and expressed in micromoles per litre
  micromoles per liter | 14.4 (9.2) | 14.2 (7.7) | 14.3 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Non-fatal Stroke, Non-fatal Myocardial Infarction or Death Due to Vascular Causes
Time Frame: The primary outcome was measured over a median follow-up period of 3.4 years (interquartile range IQR 1.0-5.5 years).
Population: Intention to treat analysis population of all patients randomised (n=8164)
Measure: Count of Participants; unit: Participants
Arm/Group | Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug) | Placebo Tablet
Number analyzed (Participants) | 4089 | 4075
Participants | 616 | 678
Statistical Analysis 1: Comparison: Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug) vs Placebo Tablet; Test type: Superiority — We used Kaplan-Meier methods to construct cumulative time-to-event curves for the two groups, with a comparison by use of the log-rank test. We used a Cox proportional hazard model analysis to control for any potential imbalance in baseline characteristics and follow-up between the two groups; p = 0.05, Log Rank; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.82 to 1.00]
Statistical Analysis 2: Comparison: Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug) vs Placebo Tablet; Test type: Superiority; p < 0.05, Regression, Cox; Analysis before adjusting for any potential imbalance in the baseline characteristics and follow-up duration between the groups; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.81 to 1.00]
Statistical Analysis 3: Comparison: Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug) vs Placebo Tablet; Test type: Superiority; p < 0.05, Regression, Cox; Analysis after adjusting for any potential imbalance in the baseline characteristics and follow-up duration between the groups; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.81 to 1.03]

ADVERSE EVENTS:
Arm/Group | Active VITATOPS Tablet (Folic Acid 2mg, B6 25mg , B12 500ug) | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 0/4089 | 0/4075
Other Adverse Events (participants affected / at risk) | 0/4089 | 0/4075

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No